CLINICAL TRIAL: NCT06090591
Title: Cardiology Research Dubrava: Single Centre, Prospective Registry
Brief Title: Cardiology Research Dubrava Prospective Registry
Acronym: CaRDr
Status: Recruiting | Type: Observational
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Ivan Zeljkovic, M.D., Ph.D., Associate Professor, University Hospital Dubrava
Other Study IDs: DUH-012017
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure; Arrhythmias, Cardiac; Atrial Fibrillation; Acute Coronary Syndrome
Keywords: chronic heart failure; acute coronary syndrome; SGLT-2 inhibitors; anticoagulants; atrial fibrillation; NTproBNP; cardiac implanted electronic device; observationl
MeSH Terms: conditions — Heart Failure; Arrhythmias, Cardiac; Atrial Fibrillation; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Acute coronary syndrome - ACS: patients who were diagnosed with acute coronary syndrome: STEMI, non-STE ACS - NSTEMI and unstable angina, who underwent coronary angiography and were prescribed with optimal medicament therapy
  Interventions: Other: SGLT-2 inh therapy, CIED implantation, thromboaspiration,
- Transcatheter aortic valve implantation - TAVI: patients with aortic stenosis who underwent transcatheter percotaneous implantation of the arteficial aortic valve
  Interventions: Other: SGLT-2 inh therapy, CIED implantation, thromboaspiration,
- Venous thromboembolism - VTE: patients with pulmonary embolism and deep vein thrombosis, with a focus on those who underwent thromboaspiration due to high or medium-high risk pulmonary embolism
  Interventions: Other: SGLT-2 inh therapy, CIED implantation, thromboaspiration,
- Heart failure with SGLT2 inhibitor therapy included - HF-SGLT2: patients with heart failure with reduced, mid-reduced and preserved systolic function who were prescribed with a SGLT-2 inhibitor therapy, and other optimal medicament therapy for HF
  Interventions: Other: SGLT-2 inh therapy, CIED implantation, thromboaspiration,
- Cardiac implantable electronic device - CIED: patients who were implanted with a cardiac implantable electronic device: pacemaker, conduction system pacing device, cardioverter-defibrilator or cardiac resynchronization therapy with or without defibrilator option
  Interventions: Other: SGLT-2 inh therapy, CIED implantation, thromboaspiration,
- Arrhythmias: patients who underwent electrophysiology study, including PVI for atrial fibrillation, as well as SVT ablations, and ventricular arrhythmia ablation (both premature ventriclar beats and ventricular tachycardia ablation in ischsmic and non-ischemic cardiomyopathy).

INTERVENTIONS:
Other: SGLT-2 inh therapy, CIED implantation, thromboaspiration, — long-term follow up and observation of patients treated in Cardiology department in the tertiary center and University hospital
  Groups: Acute coronary syndrome - ACS; Cardiac implantable electronic device - CIED; Heart failure with SGLT2 inhibitor therapy included - HF-SGLT2; Transcatheter aortic valve implantation - TAVI; Venous thromboembolism - VTE

SUMMARY:
Cardiology Research Dubrava registry is a prospective, single centre registry including patients with acute coronary syndrome with and without ST segment elevation, patients with heart failure who were prescribed with SGLT-2 inhibitors, patients implanted with TAVI, patients with venous thromboembolism, patients with pulmonary embolism who underwent thromboaspiration procedure, patients implanted with ICD, CRT and conduction system pacing devices, as well as patients with atrial fibrillation who underwent pulmonary vein isolation and are prescribed with long-term anticoagulation therapy.

DETAILED DESCRIPTION:
Cardiology Research Dubrava registry is a prospective, single centre registry including patients with acute coronary syndrome with and without ST segment elevation, patients with heart failure who were prescribed with SGLT-2 inhibitors, patients implanted with TAVI, patients with venous thromboembolism, patients with pulmonary embolism who underwent thromboaspiration procedure, patients implanted with ICD, CRT and conduction system pacing devices, as well as patients with atrial fibrillation who underwent pulmonary vein isolation and are prescribed with long-term anticoagulation therapy.

In this long-term follow-up registry we plan to collect data on clinical status, standard laboratory results including lipidogram values, NTproBNP values after specific interventions (in.ex. TAVI implantation, SGLT2inh prescripition), bleeding complications, and every major cardiovascular event, including cardiovascular death and all cause death.

ELIGIBILITY:
Inclusion Criteria: patients implanted with CIED, or with VTE, or with ACS or with TAVI -

Exclusion Criteria: non compliance, not undergoing follow-up at this center

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with different cardiology pathology and diseases including arrhythmias, heart failure, venousn thromboembolism, implanted with CIED
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2033-01 (Estimated); Study Completion 2033-06 (Estimated)

PRIMARY OUTCOMES:
cardiovascular death | 10 years
  death due to cardiovascular etiology during long term follow-up
freedom from atrial arrhythmias | 10 years
  Freedom from atrial arrhythmias after PVI during mid-term folow-up (1 year) and long-term follow-up
Time to revascularization | 10 years
  Time to revascularization during acute coronary syndrome
Bleeding complications | 10 years
  Bleeding complications during long-term follow-up in patients prescribed with oral anticoagulation and/or antithrombotic therapy
Laboratory levels of NTproBNP | 10 years
  Laboratory levels of NTproBNP in patients with AFib after PVI, in patients with HF prescribed with SGLT2 inhibitors, in patients with ACS after complete revasculariazation, in patients implanted with CIED

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Jurin, M.D., Study Chair — Dubrava University Hospital; Irzal Hadzibegovic, M.D., Principal Investigator — Dubrava University Hospital; Nikola Pavlovic, M.D., Principal Investigator — Dubrava University Hospital; Marin Pavlov, M.D., Principal Investigator — Dubrava University Hospital; Mario Udovicic, M.D., Principal Investigator — Dubrava University Hospital; Danijel Unic, M.D., Principal Investigator — Dubrava University Hospital; Ana Jordan, M.D., Principal Investigator — Dubrava University Hospital; Tomislav Sipic, M.D., Principal Investigator — Dubrava University Hospital; Diana Rudan, M.D., Principal Investigator — Dubrava University Hospital; Sime Manola, M.D., Study Director — Dubrava University Hospital
Locations (1):
- Dubrava University Hospital, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No